CLINICAL TRIAL: NCT06157359
Title: Effect of Scalp Nerve Block on the Quality of Recovery in Patients Undergoing Supratentorial Tumor Resection
Brief Title: Effect of SNB on the QoR in Patients Undergoing Supratentorial Tumor Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-0826
Record Dates: First submitted 2023-11-14; First posted 2023-12-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Analgesia; Quality of Recovery; Supratentorial Tumor; Craniotomy; Scalp Nerve Block
Keywords: Supratentorial tumor resection; Scalp nerve block; quality of recovery; postoperative analgesia
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in the control group will receive general anesthesia without the nerve blocks.
- SNB group (Experimental): Participants randomized to the SNB group will receive general anesthesia combined with SNB using 0.75% ropivacaine, which will be performed by the same attending anesthesiologist.
  Interventions: Procedure: scalp nerve block

INTERVENTIONS:
Procedure: scalp nerve block — In the SNB group, bilateral scalp nerve blocks will performed using 20 mL of 0.75% ropivacaine after anesthesia induction. To cover the area of surgical incision and skull clamp, seven scalp nerves including the supratrochlear, supraorbital, zygomaticotemporal, auriculotemporal, lesser occipital and greater occipital nerves, are blocked bilaterally by injecting 1-2 ml of the solution using a 25-gauge needle.
  Other Names: 0.75% ropivacaine
  Arms: SNB group

SUMMARY:
Patients with Supratentorial tumor undergoing craniotomy have a higher risk of postoperative pain, which will affect their postoperative quality of recovery (QoR). Although scalp nerve block (SNB) can alleviate postoperative pain, the effect on postoperative QoR in patients with supratentorial tumor undergoing craniotomy is still unclear. This study is aimed to explore the effect of SNB on postoperative QoR in this population. To explore the effect, we design a randomized controlled trial in which 84 patients with supratentorial tumor will be randomly assigned to either the SNB group or control group. The primary outcome is 15-item QoR score at 24 h after surgery. The secondary outcomes include 15-item QoR scores at 72 h after surgery, Riker Sedation-Agitation Scale, nausea and vomiting, intraoperative opioids and propofol consumption, perioperative heart rate and mean artery pressure, the duration of anesthesia and surgery, time to extubation, PACU duration, the length of postoperative days, adverse events within 72h and total medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65;
* the diagnosis was supratentorial tumor;
* scheduled for elective supratentorial craniotomy with general anesthesia ;
* the American Society of Anesthesiologists physical status I-III;

Exclusion Criteria:

* the BMI≦18kg/m2 or BMI≧30kg/m2;
* refusing to sign written informed consent;
* anticipated surgery duration is too short (<2 h) or too long (>6 h);
* liver or kidney dysfunction, severe cardiopulmonary failure or nervous system disease ;
* with other malignancies ;
* severe hematological disease and / or abnormal coagulation function;
* fever, systemic and / or scalp infection;
* tumors are metastases, aneurysms, hemangioma, or located in the skull base, or located in functional brain areas such as language and movement;
* allergy to any drug used in this study;
* a history of craniotomy tumor resection;
* preoperative usage of antiinflammatory agents or analgesics;
* pregnant women, lactating women, illiterate people, people with cognitive impairment, a history of mental illness, unable to communicate and complete the scale assessment;
* patients with severe hemodynamic disturbances or other life-threatening complications during the operation, or those transferred to the intensive care unit (ICU) after surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
the 15-item QoR score at 24 hours after surgery | up to day1 after surgery
  The quality of postoperative recovery is assessed by QoR-15 on the first day after operation.

SECONDARY OUTCOMES:
the 15-item QoR score at 72 hours after surgery | up to day3 after surgery
  The quality of postoperative recovery is assessed by QoR-15 on the third day after operation.
postoperative pain scores | up to day3 after surgery
  Pain intensity is evaluated with the numerical rating scale (0-10, 0 = no pain, 10 = unbearable pain) at 6 time points: 20 minutes after extubation, discharge from PACU, 6 hours, 12 hours, 24 hours, and 72 hours following surgery. The worst pain score during each interval is recorded.
Riker Sedation-Agitation Scale | during in PACU, an average of 3 hours
  Riker Sedation-Agitation Scale is assessed at 2 time points: 20 minutes after extubation and discharge from PACU.
nausea and vomiting | up to day3 after surgery
  Nausea and vomiting is assessed by postoperative nausea and vomiting score (0, no nausea or vomiting; 1, nausea but no vomiting; 2, vomiting once or twice; 3, vomiting on more than two occasions) at 3 time points: discharge from PACU, 24 hours, and 72 hours after operation.
opioids and propofol consumption | during operation and in PACU, an average of 8 hours
  Total drug dose of sufentanil, remifentanil and propofol consumption is recorded during operation and in PACU.
mean artery pressure and heart rate | during operation and in PACU, an average of 8 hours
  Mean artery pressure and heart rate are recorded at 6 time points: before anesthesia induction (T0), after placement of the skull clamp (T1), beginning of surgery (T2), end of surgery (T3), 20 minutes after extubation (T4) , and discharge from PACU (T5).
time to critical events | during hospitalization, an average of 10 days
  The time to critical events are recorded, including the duration of anesthesia and surgery, time to extubation, PACU duration, postoperative hospital days and so on.
adverse events | up to day3 after surgery
  Adverse events within 72 hours after operation are recorded.
total medical expenses | during hospitalization, an average of 10 days
  The total medical expenses is recorded during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated Hospital School of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No